CLINICAL TRIAL: NCT02153502
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deuterium Modified Dextromethorphan Hydrobromide/Quinidine Sulfate) as an Adjunctive Therapy in Patients With Major Depressive Disorder With an Inadequate Response to Antidepressant Treatment
Brief Title: Efficacy, Safety, and Tolerability Study of AVP-786 as an Adjunctive Therapy in Patients With Major Depressive Disorder With an Inadequate Response to Antidepressant Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-AVP-786-201
Record Dates: First submitted 2014-05-29; First posted 2014-06-03 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVP-786 (Experimental)
  Interventions: Drug: AVP-786 (d6-dextromethorphan hydrobromide and quinidine sulfate combination)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVP-786 (d6-dextromethorphan hydrobromide and quinidine sulfate combination) — AVP-786 capsules administered twice a day over a 10-week period
  Arms: AVP-786
Drug: Placebo — Placebo capsules administered twice a day over a 10-week period
  Arms: Placebo

SUMMARY:
The objectives of this 10-week study are to evaluate the efficacy, safety, and tolerability of AVP 786 as an adjunctive therapy compared with placebo in patients with major depressive disorder (MDD) who have shown an inadequate response to standard antidepressant treatment. A secondary objective of this study is to assess the pharmacokinetics (PK) of AVP-786 and potential correlations with pharmacodynamic effects.

DETAILED DESCRIPTION:
It is estimated that up to approximately 200 patients will participate in the study at approximately 30 enrolling centers in the US.

Eligible patients for this study must have MDD as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria, and have shown an inadequate response to standard antidepressant treatment.

This is a multicenter, randomized, double-blind, placebo-controlled, study of 10 weeks duration.

Following screening procedures for assessment of inclusion and exclusion criteria, eligible patients will be randomized into the study. Study medication will be administered orally twice a day (BID) (1 capsule in the morning and 1 capsule in the evening, approximately 12 hours apart) throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depressive episode ≤ 24 months in duration
* HAM-D17 score ≥ 20.
* Documented to not have a significant (25% or greater) change in QIDS-SR16 score between Screening and Baseline visits.
* Patients have been deemed to have an inadequate response (less than 50% symptom reduction) to at least 1 but no more than 3 adequate antidepressant trials during the current depressive episode.
* Patients must be receiving ongoing treatment with an adequate dose of antidepressants.
* Body Mass Index (BMI) of 18-35 kg/m².

Exclusion Criteria:

* History of myasthenia gravis.
* Have cardiovascular concerns such as:

  * History of complete heart block, QT interval corrected for heart rate (QTc) prolongation, or torsades de pointes.
  * QTc using the Fridericia's formula (QTcF) at screening > 450 msec for males and > 470 msec for females based on central review at the screening visit, unless due to ventricular pacing.
  * Any family history of congenital QT interval prolongation syndrome.
* Known hypersensitivity/intolerance to DM, Q, opiate drugs (codeine, etc.), or any other ingredient of the study medication.
* Pose a current suicide risk, as evidenced by any of the following:

  * It is the judgment of the investigator that the subject may be at risk for suicide.
  * The subject is rated a "yes" to question 4 or question 5 on the Baseline C-SSRS, if the most recent episode occurred within the past 12 months.
  * The subject has attempted suicide within the past 6 months
* Presence of any other current DSM-IV-TR Axis I disorders with the exception of: generalized anxiety disorder (GAD: 300.02), social anxiety disorder (300.23), dysthymic disorder (300.4), or specific phobia (300.29). Patients with co-morbid GAD, social anxiety disorder, or specific phobia are ineligible if the co-morbid condition is clinically unstable, or has been the primary focus of treatment within the 6 month period prior to screening
* Axis I diagnosis of:

  * Delirium, dementia, amnestic, or other cognitive disorder;
  * Schizophrenia or other psychotic disorder, based on the M.I.N.I.;
  * Bipolar I or II disorder, based on the M.I.N.I.
* Clinically significant Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Montgomery-Ǻsberg Depression Rating Scale (MADRS) total score | Visit 5 (Day 70) Week 10
  Montgomery-Ǻsberg Depression Rating Scale (MADRS) total score in patients receiving AVP 786 compared with patients administered placebo

SECONDARY OUTCOMES:
17-item Hamilton Rating Scale for Depression (HAM-D17) | Visit 5 (Day 70) Week 10
Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH ATRQ) | Visit 5 (Day 70) Week 10
16-item Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR16) | Visit 5 (Day 70) Week 10
Sheehan Disability Scale (SDS) | Visit 5 (Day 70) Week 10
Clinical Global Impression of Severity of Illness (CGI-S) | Visit 5 (Day 70) Week 10
Clinical Global Impression of Change (CGI-C) | Visit 5 (Day 70) Week 10
EuroQOL 5 Dimension 5 Level (EQ-5D-5L) | Visit 5 (Day 70) Week 10
Patient Global Impression of Change (PGIC) | Visit 5 (Day 70) Week 10
7-item Generalized Anxiety Disorder (GAD-7) | Visit 5 (Day 70) Week 10

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Birmingham, Alabama
  - Bellflower, California
  - Costa Mesa, California
  - Garden Grove, California
  - Lomita, California
  - Oceanside, California
  - Riverside, California
  - Santa Ana, California
  - Sherman Oaks, California
  - Denver, Colorado
  - Bradenton, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Decatur, Georgia
  - Hoffman Estates, Illinois
  - Valparaiso, Indiana
  - Baltimore, Maryland
  - Glen Burnie, Maryland
  - Boston, Massachusetts
  - Brooklyn, New York
  - New York, New York
  - Staten Island, New York
  - Garfield Heights, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Murray, Utah